CLINICAL TRIAL: NCT00776048
Title: The Validation of a New Method to Evaluate the Effects of Chemoneurolytic Intervention on Balance and Community Ambulation in Spastic Hemiplegic Patients
Brief Title: Validation of an Obstacle Course Used in Patients With Muscle Tightness
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kessler Foundation (Other)
Responsible Party: Elie Elovic, M.D., Kessler Medical Rehabilitation Research and Education Center
Other Study IDs: E56806
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2008-10

CONDITIONS: Stroke; Traumatic Brain Injury; Multiple Sclerosis; Spasticity; Healthy Controls
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ABI: Acquired brain injury with lower limb spasticity
- Healthy Controls: Age matched healthy controls

SUMMARY:
This study is being conducted to compare healthy patients versus patients with muscle tightness in their leg(s) after an acquired brain injury using walking trials time, a balance test, and foot pressure data. This data is obtained using foot pressure sensors, timers, and distance walked.

DETAILED DESCRIPTION:
This study is being conducted to demonstrate the objective utility of the use of pedobarography as a tool to differentiate normal controls from people with spastic gait as well as having utility in objectification of treatment effect on level surfaces and on a ADA based obstacle course.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Must wear shoe size 5½ - 11 US womens or size 6 - 13 US mens
* For treatment group be a clinical patient being treated for lower extremity spasticity

Exclusion Criteria:

* Age matched controls must have no significant neurological or orthopedic disease that would effect their gait
* Clinical patients who are unable to walk for 1 minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects ages > 18 years of age for this study. A total of up to 10 age matched controls and 30 clinical patients with lower extremity spasticity will be enrolled. Of the 30 clinical patients, 20 clinical patients will have received BOTOX ® injections from their clinical physician after their first visit.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the objective utility of the use of pedobarography to differentiate normal controls from people with spastic gait as well as having utility in objectification of treatment effect on level surfaces and on a ADA based obstacle course. | 4 months post acquired brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Elie P Elovic, M.D., Principal Investigator — Kessler Foundation
Locations (1):
- KesslerMRREC, West Orange, New Jersey, United States

REFERENCES:
- See also: KesslerMRREC Traumatic Brain Injury Website — https://kesslerfoundation.org/research/nnjtbis/